CLINICAL TRIAL: NCT06823583
Title: Multi-Site Feasibility Testing of the Ventricular Assist Device Anticipatory Guidance Tool
Status: Recruiting | Type: Observational
Sponsor: Bryan Heart (Other)
Collaborators: International Consortium of Circulatory Assist Clinicians (Other); International Society for Heart and Lung Transplantation (Other)
Responsible Party: Principal Investigator, Sarah E Schroeder, Left Ventricular Assist Device Nurse Practitioner and Program Manager, Bryan Heart
Other Study IDs: MCS-VAD-003
Record Dates: First submitted 2025-01-12; First posted 2025-02-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Ventricular Assist Device; Advanced Heart Failure; Anticipatory Guidance
Keywords: expectations; VAD; Advanced Heart Failure; Anticipatory Guidance; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- VAD Clinician Cohort: Up to four VAD Clinicians at each of the three participating sites (a maximum total of 12) will provide feedback and evaluation of the VAD AG Tool v5.0 following consenting.
- VAD Patient Cohort: Each of the three sites will enroll a minimum of 3 patients and no more than 5 potential VAD patients (total of 21 for the three sites) to provide evaluation and feedback of accuracy and feasibility of the VAD AG Tool v5.0, occurring at 3-, 6- and 12-months following VAD implant. All patient participants following consenting, will receive the tool pre-surgery and provide evaluation and guidance post surgery, along with de-identifiable demographic and clinic data.

SUMMARY:
There are a variety of educational documents available to help in a participant's decision for VAD implant, however there is little information available to potential participants to help understand areas of satisfaction and concern following a VAD implant as various time points. The investigators want to provide better patient care through increased education and awareness beyond surgical outcomes and contribute to patient understanding of "what to expect" following a VAD implant.

The investigators have created an anticipatory guidance (AG) tool based upon previous responses recorded in a local program's database, from the Quality of Life with a Left Ventricular Assist Device (QoLVAD) questionnaire. This questionnaire has five different domains (physical, social, emotional, cognitive thinking and spiritual/well-being). Investigators have previously analyzed responses to determine common areas of satisfaction and concern at 3-, 6-, 12- and 24-months post-VAD implant to better understand quality of life when living with a VAD. Investigators have had both VAD clinicians and VAD patients initially evaluate the tool to determine accuracy and effectiveness of the anticipatory guidance (AG) tool.

DETAILED DESCRIPTION:
Advanced heart failure (HF) accounts for up to 10% of the overall HF population, and is demonstrated through increased hospitalizations, worsening shortness of breath and decrease in energy. A left ventricular assist device (VAD) and/or cardiac transplantation are promising surgical options to treat advanced HF beyond traditional guideline driven medical therapy, however not always designed for everyone. There are extensive educational materials available preoperatively designed to provide additional information to ease the decision-making process when receiving a VAD, yet most of this material is used to help decide on whether to get a VAD and has less to do with what to expect following a VAD. No information exists to date on describing expectations and outcomes at various time points following VAD. Anticipatory guidance (AG) models primarily exist in the pediatric populations to help parents and caregivers understand the "typical" milestones of what to expect. There are scarce AG models available for adults with chronic comorbid conditions, such as HF. An AG tool specific to VAD patients would be beneficial as preoperative education for potential VAD patients to help better understand the more commonly defined expectations of outcomes beyond adverse event risks, and in turn, hopefully decreases anxiety and depression post-VAD implant, improve domains of health-related quality of life (HRQoL), and decrease hospitalizations.

The Phase 1 study evaluated the development of a prototype AG tool from both longitudinal data analyzed from internal "Quality of Life with a Left Ventricular Assist Device" (QoLVAD) questionnaires that were previously completed as part of a local program's database, and from additional supporting literature. The prototype AG tool has undergone a two-part Delphi method evaluation by 10 international VAD clinicians, and necessary modifications were made based upon results from the two-part Delphi method. An additional round of Delphi method evaluation with local VAD patients was completed with final modifications to reflect the responses from the VAD patients to develop the "VAD AG Tool v5.0". The Phase 2 tool will be referred to as the "VAD AG tool v5.0".

For this phase 2 study, the purpose is to evaluate the VAD AG tool v5.0 across three VAD implanting centers in the United States, with the perspectives of both VAD patients and clinicians. This will be accomplished through four aims: 1. Evaluate clinician perspectives of the VAD AG Tool v5.0; 2. Preoperative distribution of the VAD AG tool v5.0 for consented participants across three VAD implanting centers, to read preoperatively, and evaluate at postoperative time points (3, 6 and 12-months); 3. Describe postoperative VAD patient perceptions of VAD AG tool v5.0 at three time points (3, 6, and 12-months); and 4. Evaluate relationships between HRQoL and the following: anxiety, depression, cognition, and hospital readmissions.

ELIGIBILITY:
Inclusion Criteria:

(For patient inclusion):

* scheduled for a VAD implantation
* English-speaking as the VAD AG Tool v5.0 has not yet been translated beyond English age ≥19 years at the time of implant as most states in North America have an age of majority for consent signing.

(-VAD clinician for the clinician evaluation process)

Exclusion Criteria:

* Not scheduled for VAD surgery
* Non English speaking
* <19 yrs of age (Not a VAD Clinician for the clinician evaluation process)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced heart failure patients will be approached by their internal VAD teams who have been scheduled for a VAD implantation. Only age requirement is >/= 19 as the age of majority in most states for consenting is 19. The goal is to consent consecutively so as to limit selection bias as much as able to. This is a feasibility study so consecutive approaching is key.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-08-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinician perspectives | First two weeks of study initiation.
  Evaluate clinician perspectives of the Ventricular Assist Device Anticipatory Guidance Tool (VAD AG Tool) v5.0 for accuracy, by completing an evaluation where each item will be scored 1-4, as follows: 1 Not Relevant, 2 Somewhat Relevant, 3 Quite Relevant, 4 Highly Relevant

OTHER OUTCOMES:
Distribution of the Ventricular Assist Device Anticipatory Guidance Tool (VAD AG Tool) v5.0 | 12 months
  Each site investigator will validate that the Ventricular Assist Device Anticipatory Guidance Tool (VAD AG Tool) v5.0 was preoperatively distributed.
Postoperative patient perceptions of Ventricular Assist Device Anticipatory Guidance Tool (VAD AG Tool) v5.0 | 12 months
  Consented patients will provide prospectives of the Ventricular Assist Device Anticipatory Guidance Tool (VAD AG Tool) v5.0, through a patient evaluation form where all tool items will be scored on a 1-4 scale, where 1 is Not Important, 2 is Somewhat Important, 3 is Quite Important, 4 is Highly Important
Complete post-operative Quality of Life with a Left Ventricular Assist Device (QoLVAD) | 12 months
  All consented participants will complete the QoLVAD questionnaire at three time points (3-6-12 months)
Complete post-operative Generalized Anxiety Disorder 7-item scale at three different time points | 12 months
  All consented participants will complete the GAD-7 assessment at three time points (3-6-12 months)
Complete post-operative Patient Health Questionnaire-9 tool at three different time points | 12 months
  All consented participants will complete the PHQ-9 assessment at three time points (3-6-12 months)
Complete post-operative Trailmaking B assessment at three different time points | 12 months
  All consented participants will complete the Trailmaking B assessment at three time points (3-6-12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Mathue Baker, MD, Study Chair — Bryan Heart
Locations (2):
- United States (2):
  - Bryan Heart, Lincoln, Nebraska
  - Advocate Aurora Health, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Each participant will have de-identifiable demographic and clinical data gathered for the purposes of this study, along with the data obtained from each pre-VAD questionnaire will be gathered by each site PI and provided to the primary study PI. The de-identifiable demographic and clinical data will be entered on the Pre- or Post-operative Data Collection Forms, and copies will be sent directly to the primary study PI. All de-identifiable study data will be stored in a password protected computer at Bryan Heart, located in the primary study PI's Mechanical Circulatory Support office. All data (which will be de-identified) will only be accessible directly by the primary study PI and the co-investigators. No direct identifiable individualized participant data will be shared with the primary study PI or co-investigators as all data that is to be sent will be coded with the site number, the sequence in consenting and the interval form number.
Supporting Information: SAP
Time Frame: August 2025 is the expected start date, and the goal is to have all data collected and back to the primary study PI by November to December 2026 to which no additional data will need to be collected once the 12-month data collection has been completed.
Access Criteria: All Individualized Patient Data will be de-identifiable. The primary study PI will be the organizer of all data and then once put all together, the primary study PI will share the data with the additional co-investigators. No other identifying information will be provided as all patients will have a specific code (site # (1-4), sequence of consenting (1-7) and lettering of interval (A-preop, B-3months, C-6months or D-12months). All data will be kept in a password protected desktop used solely by the primary study PI in Bryan Heart Mechanical Circulatory Support office to which the data is protected through Bryan Heart's IT department policies.

REFERENCES:
- [Background] Waldenburger N, Steinecke M, Peters L, Junemann F, Bara C, Zimmermann T. Depression, anxiety, fear of progression, and emotional arousal in couples after left ventricular assist device implantation. ESC Heart Fail. 2020 Oct;7(5):3022-3028. doi: 10.1002/ehf2.12927. Epub 2020 Jul 28. PMID 32725771
- [Background] Highs and Lows of Life with a Left Ventricular Assist Device: Multi-Dimensional Perspectives Schroeder, S.E. et al. The Journal of Heart and Lung Transplantation, Volume 43, Issue 4, S606
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Longitudinal Quality of Life Assessment Following Ventricular Assist Device Therapy: A Pilot Study Using the QOLVAD Questionnaire Schroeder, S.E. et al. The Journal of Heart and Lung Transplantation, Volume 39, Issue 4, S91
- [Background] Sandau KE, Lee CS, Faulkner KM, Pozehl B, Eckman P, Garberich R, Weaver CE, Joseph SM, Hall S, Carey SA, Chaudhry SP, Schroeder SE, Hoffman RO 3rd, Feldman D, Birati EY, Soni M, Marble JF, Jurgens CY, Hoglund B, Cowger JA. Health-Related Quality of Life in Patients With a Left Ventricular Assist Device (QOLVAD) Questionnaire: Initial Psychometrics of a New Instrument. J Cardiovasc Nurs. 2021 Mar-Apr 01;36(2):172-184. doi: 10.1097/JCN.0000000000000774. PMID 33306621
- [Background] Birriel B, Alonso W, Kitko LA, Hupcey JE. Family caregiver-reported outcomes regarding decision-making for left ventricular assist device implantation. Heart Lung. 2019 Jul-Aug;48(4):308-312. doi: 10.1016/j.hrtlng.2019.03.002. Epub 2019 Apr 10. PMID 30981423
- [Background] Kitko LA, Hupcey JE, Birriel B, Alonso W. Patients' decision making process and expectations of a left ventricular assist device pre and post implantation. Heart Lung. 2016 Mar-Apr;45(2):95-9. doi: 10.1016/j.hrtlng.2015.12.003. Epub 2015 Dec 29. PMID 26742707
- [Background] McIlvennan CK, Magid KH, Ambardekar AV, Thompson JS, Matlock DD, Allen LA. Clinical outcomes after continuous-flow left ventricular assist device: a systematic review. Circ Heart Fail. 2014 Nov;7(6):1003-13. doi: 10.1161/CIRCHEARTFAILURE.114.001391. Epub 2014 Oct 7. PMID 25294625
- [Background] Sandau KE, Hoglund BA, Weaver CE, Boisjolie C, Feldman D. A conceptual definition of quality of life with a left ventricular assist device: results from a qualitative study. Heart Lung. 2014 Jan-Feb;43(1):32-40. doi: 10.1016/j.hrtlng.2013.09.004. Epub 2013 Oct 2. PMID 24239297
- [Background] Mehra MR, Goldstein DJ, Cleveland JC, Cowger JA, Hall S, Salerno CT, Naka Y, Horstmanshof D, Chuang J, Wang A, Uriel N. Five-Year Outcomes in Patients With Fully Magnetically Levitated vs Axial-Flow Left Ventricular Assist Devices in the MOMENTUM 3 Randomized Trial. JAMA. 2022 Sep 27;328(12):1233-1242. doi: 10.1001/jama.2022.16197. PMID 36074476
- [Background] Bytyci I, Bajraktari G. Mortality in heart failure patients. Anatol J Cardiol. 2015 Jan;15(1):63-8. doi: 10.5152/akd.2014.5731. Epub 2014 Aug 19. PMID 25550250